CLINICAL TRIAL: NCT02852356
Title: Prospective Observational and Validation Study Using Time-lapse Morphometry MIRI Imaging Incubator (TiMMI Study)
Brief Title: Validation Study Using a Time-lapse Morphometry MIRI Imaging Incubator
Acronym: TiMMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ovation Fertility (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2016-TiMMI-001
Record Dates: First submitted 2016-07-28; First posted 2016-08-02 (Estimated); Results first posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-04

CONDITIONS: Fertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control Incubator (No Intervention): Standard Incubator
- MIRI-TL Timelapse Incubator (Experimental): Timelapse incubator
  Interventions: Device: MIRI-TL Incubator
- Culture Coin Dish (Experimental): Culture Coin dish for embryo culture
  Interventions: Device: MIRI-TL Incubator
- Control dish (No Intervention): Control Dish for embryo culture

INTERVENTIONS:
Device: MIRI-TL Incubator — MIRI-TL Timelapse incubator
  Arms: Culture Coin Dish; MIRI-TL Timelapse Incubator

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the MIRI-TL time-lapse incubator and CultureCoin dish compared to standard big-box incubators and standard culture dishes used for embryo culture.

DETAILED DESCRIPTION:
Following randomization and standard ovarian stimulation protocols to obtain a sufficient number of mature (MII) oocytes, these oocytes will be fertilized by Intra-Cytoplasmic Sperm Injection (ICSI). If a patient has been randomized to the study group, all inseminated oocytes and subsequently all fertilized diploid (2PN) zygotes will be placed in the CultureCoin and then into the MIRI-TL Time-lapse incubator and cultured as per normal protocol to the blastocyst stage (Day 5/6 or 7). Top quality blastocyst(s) will be transferred and monitored for implantation, pregnancy and ongoing birth. Embryo transfers will either occur in a fresh or frozen embryo transfer cycle.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Women undergoing in vitro fertilization treatment using their own or frozen oocytes
* Fresh or Frozen Embryo Transfer
* Fertilization by ICSI
* At least 4 diploid (2PN) embryos at fertilization check
* Willing to have all inseminated oocytes imaged by Miri
* Willing to comply with study protocol and procedures Willing to provide written informed consent

Exclusion Criteria:

* Fertilization using surgically removed sperm
* History of cancer

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2016-07; Primary Completion 2017-12-22 (Actual); Study Completion 2017-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew VerMilyea, PhD, Principal Investigator — Ovation Fertility
Locations (1):
- Ovation Fertility, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Non-identified data regarding embryo development and pregnancy outcomes may be shared and discussed through presentations and publications.
Time Frame: Project has ceased
Access Criteria: Project has ceased

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Incubator | MIRI-TL Timelapse Incubator | Culture Coin Dish | Control Dish
Started | 31 | 31 | 0 | 0
Completed | 31 | 31 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: patients in the dishes equal number in incubator
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Incubator | MIRI-TL Timelapse Incubator | Culture Coin Dish | Control Dish | Total
Number analyzed (Participants) | 31 | 31 | 0 | 0 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 |  |  | 0
  Between 18 and 65 years | 31 | 31 |  |  | 62
  >=65 years | 0 | 0 |  |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 31 |  |  | 62
  Male | 0 | 0 |  |  | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Positive bHCG Level as Detected by a Blood Test
Description: Human Chorionic Gonadotropin (hormone made by cells formed in the placenta) are detected by a blood test. An hCG level >50mIU/mL is considered to be a successful pregnancy.
Time Frame: 14 days after embryo transfer
Population: number in incubator equals number in dish
Measure: Number; unit: Participants
Arm/Group | Control Incubator | MIRI-TL Timelapse Incubator | Culture Coin Dish | Control Dish
Number analyzed (Participants) | 31 | 31 | 0 | 0
Participants | 19 | 19 |  |

2. Secondary Outcome: Number of Patients With Embryo Implantation
Description: Presence of Gestational Sac by ultrasound indicates a positive pregnancy.
Time Frame: 28 days
Population: number in incubator equals number in dish
Measure: Number; unit: Participants
Arm/Group | Control Incubator | MIRI-TL Timelapse Incubator | Culture Coin Dish | Control Dish
Number analyzed (Participants) | 31 | 31 | 0 | 0
Participants | 15 | 14 |  |

3. Secondary Outcome: Embryo Development
Description: Blastocyst Utilisation Rate (number of fertilised embryos which develop to usable blastocysts)
Time Frame: 7 days
Population: number in incubator equals number in dish
Measure: Count of Units; unit: Embryos
Units Other Than Participants: Embryos
Arm/Group | Control Incubator | MIRI-TL Timelapse Incubator | Culture Coin Dish | Control Dish
Number analyzed (Participants) | 31 | 31 | 0 | 0
Number analyzed (Embryos) | 150 | 165 | 0 | 0
Embryos | 52 | 54 |  |

4. Post Hoc Outcome: Number of Patients With Live Birth
Description: Reported live birth of a child
Time Frame: 9 months
Population: No participants in the culture coin Dish or the control dish.
Measure: Number; unit: participants
Arm/Group | Control Incubator | MIRI-TL Timelapse Incubator | Culture Coin Dish | Control Dish
Number analyzed (Participants) | 31 | 31 | 0 | 0
participants | 10 | 9 |  |

ADVERSE EVENTS:
Time Frame: 9 months
Description: No adverse events were reported in this study. All-Cause Mortality was not monitored/assessed.
Arm/Group | Control Incubator | MIRI-TL Timelapse Incubator | Culture Coin Dish | Control Dish
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/31 | 0/31 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-06-15): https://cdn.clinicaltrials.gov/large-docs/56/NCT02852356/Prot_SAP_000.pdf
  • Informed Consent Form (2016-06-15): https://cdn.clinicaltrials.gov/large-docs/56/NCT02852356/ICF_001.pdf